CLINICAL TRIAL: NCT06206785
Title: Resting Energy Expenditure in Palliative Cancer Patients (REPAT) - an Explorative Study in Patients With Incurable Cancer
Brief Title: Resting Energy Expenditure in Palliative Cancer Patients
Acronym: REPAT
Status: Recruiting | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); UiT The Arctic University of Norway (Other)
Responsible Party: Sponsor
Other Study IDs: 622545
Record Dates: First submitted 2023-12-14; First posted 2024-01-16 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Cachexia
MeSH Terms: conditions — Neoplasms; Cachexia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study purpose is to measure REE by indirect calorimetry and to determine limits of agreement with confidence intervals between measured REE and predictive equations for determination of energy requirements in patients with incurable cancer. Clinical factors associated with hyper- and hypometabolism will be elucidated. Data will be obtained from patient journals in combination with measurements of REE and registration of survival. Data will be collected at one timepoint and survival will be monitored prospectively.

ELIGIBILITY:
Inclusion Criteria:

* A verified diagnosis of an incurable malignant disease
* Hospitalized at the Cancer clinic, St. Olavs Hospital
* ≥ 18 years of age
* Able to provide written informed consent
* Able to comply with all study procedures

Exclusion Criteria:

* Cognitive impairment
* In need of supplementary oxygen
* Receiving invasive or noninvasive ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is patients diagnosed with an incurable malignant disease and hospitalized at the cancer clinic, St. Olavs Hospital in the period from september 2023 to june 2026. They have to be 18 years or older and able to provide written informed consent and comply with all study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of resting energy expenditure (REE) in patients with incurable cancer measured with the COSMED Q-NRG+ Indirect Calorimeter with a Canopy Hood. | Throughout study completion, approximately 3 years.
  Investigate the agreement between the most used energy expenditure prediction equation (Harris-Benedict calculation for resting energy expenditure based on weight, height and gender) and measured REE (kilocalories/day) by indirect calorimetry in patients with incurable cancer.

SECONDARY OUTCOMES:
Clinical factors associated with hyper- and hypometabolism | Throughout study completion, approximately 3 years.
  Explore the association between patients identified as hyper-or hypometabolic (REE > 10% or < 10% of the predicted BMR (in kilocalories per day)) and a set of explanatory variables such as cancer diagnosis (type), weight loss last six months ((current/past weight)*100), symptom score (Edmonton Symptom Assessment System (ESAS)), degree of inflammation (CRP in mg/L), and survival (days after REE measurement).

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Clinic, St. Olavs Hospital, Trondheim University Hospital, Trondheim, Norway

REFERENCES:
- See also: Current Research Information System in Norway — https://app.cristin.no/projects/show.jsf?id=2636691